CLINICAL TRIAL: NCT05683249
Title: Clinical Trial to Evaluate the Safety and Efficacy of NRCT-101SR in Adult Attention Deficit Hyperactivity Disorder
Brief Title: Study to Evaluate NRCT-101SR in Adult Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Neurocentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC-018
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, parallel-arm design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRCT-101SR (Experimental): Two-tiered fixed dose of 1,500 or 2,000 mg/day. Two NRCT-101SR tablets (375 mg or 500 mg based on lean body mass) by mouth twice daily
  Interventions: Drug: NRCT-101-SR
- Matching Placebo (Placebo Comparator): Two-tiered fixed dose of 1,500 or 2,000 mg/day. Two NRCT-101SR placebo tablets (375 mg or 500 mg based on lean body mass) by mouth twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NRCT-101-SR — NRCT-101SR is a sustained release formulation. Subjects ≥ 50 kg LBM receive a total of four 500 mg tablets/day and subjects < 50kg LBM receive a total of four 375 mg tablets per day.
  Arms: NRCT-101SR
Drug: Placebo — Matching placebo
  Arms: Matching Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of NRCT-101SR compared to placebo in adult patients with ADHD aged 18 years and older.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-arm design, laboratory classroom (LC) trial to assess the efficacy and safety of NRCT-101SR compared to inactive placebo for the treatment of ADHD in adults aged 18 years and older.

After Screening, Orientation, and Baseline evaluations are complete, eligible subjects will be randomized into one of two groups (1:1) to receive NRCT-101SR or matching placebo orally twice daily, in the morning and evening, beginning the day after the Baseline visit for 6 weeks. Subjects will receive a fixed dose of 1,500 or 2,000 mg/day, based on lean body mass, split evenly between the morning and evening dosing.

Total subject participation in the study is up to approximately 13 weeks, including a screening period (up to 6 weeks), a 6-week treatment period, and an approximate 1-week follow-up period. Within 8 days prior to Baseline LC visit, subjects will complete an LC Orientation Visit. LC visits will be repeated at Week 3 and Week 6.

The primary outcome measures of the study include Permanent Product Measure of Performance (PERMP) Math Tests (number of correctly answered problems; PERMP-C) and ADHD Investigator Symptom Rating Scale (AISRS). At Baseline, Week 3 visit, and Week 6 visit, serial PERMP Math Tests at pre-dose and at 2, 4, 6, 8, 10, and 12 hours post-dose, and AISRS will be administered. LC visits will be repeated at Week 3 and Week 6. Secondary and exploratory assessments will also be conducted at the Baseline, Week 3, and Week 6 LC visits. A clinic visit will be conducted at Week 1. Pharmacokinetic (PK) sampling will be collected at the Week 3 LC visit. Safety assessments (concomitant medications, adverse events, and suicide risk) will be conducted at all clinic and remote visits/phone calls (Week 5, and follow-up); safety labs will be conducted at screening, Week 3, and Week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age at screening
2. Has a primary diagnosis of ADHD according to the Diagnostic and Statistical Manual, Fifth Edition (DSM-5) classification, confirmed with Mini International Neuropsychiatric Interview (MINI) using DSM-5 probes
3. AISRS ≥ 26 at screening and baseline, and does not change by more than 25% from screening to baseline, except subjects who stop taking ADHD medication after screening may have an increase of more than 25%
4. Has a minimum score of 4 on the CGI-S at baseline
5. Must be fluent in English, and capable of reading, writing, and communicating effectively with others and willing to participate in laboratory classroom
6. Completion of at least 10 years of formal education
7. Hearing and Vision ability sufficient to complete cognitive testing, in investigator's opinion
8. Willing and able to give informed consent
9. Total Body weight (bw) must be ≥ 50 kg and ≤ 105 kg and lean body mass (LBM) must be ≤ 75 kg at screening
10. Naïve to stimulant or non-stimulant medications used for the treatment of ADHD or have discontinued stimulants at least 2 weeks and non-stimulants at least 3 weeks prior to randomization

    Exclusion Criteria:
11. Subject is functioning below an age-appropriate level intellectually, as judged by the investigator.
12. Lifetime history of severe psychiatric symptoms of major depression requiring hospitalization, bipolar disorder, schizophrenia of schizoaffective disorder, hallucinations, or delusions. Severe comorbid disorders such as PTSD, severe obsessive-compulsive disorder, or other symptomatic presentation that, in the opinion of the examining physician, will contraindicate NRCT-101SR treatment or confound efficacy or safety assessments. Subjects with mild to moderate forms of social phobia or dysthymia, for instance, may be included.
13. History of seizures (other than infantile febrile seizures), any tic disorder (except transient tic disorder and subject has no episodes for at least 1 year), or a current diagnosis of Tourette's Disorder.
14. Recent history (within the past 1 year) of suspected substance abuse or dependence disorder (excluding stable nicotine use) in accordance with DSM-5 criteria. (Note: subject's average nicotine use should not be exceeded during each LC visit)
15. Current abnormal thyroid function as defined as abnormal screening thyroid stimulating hormone. Treatment for at least 3 months with a stable dose of thyroid medication is permitted.
16. Poor kidney function; corrected estimated glomerular filtration rate (eGFRcorr) < 40 mL/min/m2
17. History of significant gastrointestinal disorders, such as chronic diarrhea, irritable bowel syndrome, ulcerative colitis, Crohn's disease, etc.
18. Female subjects who are pregnant and/or lactating
19. A "yes" answer to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment at screening (in the past 12 months).
20. Has history of severe drug allergy or hypersensitivity to the study medication or its excipients.
21. Hypermagnesemia; magnesium > 2.5 mg/dL
22. Reproduction:

    a. Females of childbearing potential (FOCP) must be either sexually inactive abstinent) or, if sexually active, must agree to use one of the following acceptable birth control methods beginning 30 days prior to the first dose of study drug and throughout the study: i. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to first study drug administration ii. Surgically sterile male partner iii. Simultaneous use of male condom and diaphragm with spermicide iv. Established hormonal contraceptive b. Males must: i. Use 2 methods of contraception in combination if his female partner is of childbearing potential; this combination of contraceptive methods must be used from the Baseline Visit to ≥ 1 month after the last dose of study drug, or ii. Have been surgically sterilized prior to the Screening Visit.
23. Is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to the Screening Visit.
24. Currently living in an institutional facility such as a nursing home
25. Severe physical disability not associated with cognitive function that limits ability to complete testing (e.g., severe tremor, debilitating arthritis, etc.)
26. Known history of symptomatic cardiac disease, advanced atherosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke or other serious cardiac problems.
27. Known family history of sudden cardiac death or ventricular arrhythmia.
28. Serious or unstable clinically important systemic illness or disease that, in the judgment of the investigator, is likely to affect cognitive assessment, deteriorate, or affect the subject's safety or ability to complete the study, including hepatic (e.g., Child-Pugh grade C), renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, infectious, or hematologic disorders
29. Has previously participated in a NRCT-101SR investigational study or a study that includes the active ingredient of NRCT-101SR
30. Investigators and their immediate family members are not permitted to participate in the study.
31. Consumes more than a weekly average of: 2 drinks / day or more than 3 drinks in any day for males; 1 drink / day or more than 2 drinks in any day for females
32. Changes in medications or doses of medication as follows:

    1. All allowed concomitant medications, supplements, or other substances must be at stable doses for at least 30 days prior to screening and must be kept as stable as medically possible during the trial. For allowed concomitant medications, any dosing change within 30 days of Screening may be allowed if, in the opinion of the investigator, it will not affect or influence study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guosong Liu, M.D., Ph.D., Study Director — Neurocentria, Inc.
Locations (9):
- United States (9):
  - Collaborative Neuroscience Network, Garden Grove, California
  - Accel Research Sites, Lakeland, Florida
  - Accel Research Sites, Maitland, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Velocity Clinical Research - Meridian, Meridian, Idaho
  - Alcanza Clinical Research Company, Boston, Massachusetts
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Coastal Carolina Research Center - North Charleston, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 sites in the United States from 25Feb2023 to 17Jan2024.
Pre-assignment Details: A total of 223 participants were enrolled in this study. Participants were randomly assigned to 1 of 2 groups to receive NRCT-101SR or placebo for a 6-week treatment period.
Period: Overall Study
Arm/Group | NRCT-101SR | Placebo
Started | 109 | 114
Received at Least 1 Dose of Study Drug | 108 | 114
Completed | 83 | 93
Not Completed | 26 | 21
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Non-compliance with Study Drug | 2 | 0
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Two-tiered fixed dose of 1,500 or 2,000 mg/day. Two NRCT-101SR placebo tablets (375 mg or 500 mg based on lean body mass) by mouth twice daily
- Total: Total of all reporting groups
Arm/Group | NRCT-101SR | Placebo | Total
Number analyzed (Participants) | 108 | 114 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (14.07) | 36.8 (14.89) | 37.7 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 115
  Male | 53 | 54 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 77 | 85 | 162
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 11 | 26
  White | 76 | 91 | 167
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Permanent Product Measure of Performance (PERMP) - Number of Math Problems Answered Correctly (PERMP-C)
Description: PERMP is a skill adjusted math test. PERMP-C is the number of math problems answered correctly in a 10-minute session and typically ranges from 0-400 with higher scores indicating better performance. The mean of the post-dose timepoint scores will be used for evaluation.
Time Frame: Baseline and Week 6
Population: Per Protocol Population: all subjects in the mITT population who did not incur a protocol violation that impacted the efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 81 | 89
score on a scale | 21.8 (2.17) | 18.9 (2.03)

2. Primary Outcome: Change From Baseline in ADHD Investigator Symptom Rating Scale (AISRS)
Description: AISRS consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with a total score ranging from 0 to 54. Lower scores indicate less severe symptoms.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 81 | 89
score on a scale | -12.0 (1.24) | -10.7 (1.19)

3. Secondary Outcome: Change From Baseline Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A)
Description: The BRIEF-A is a standardized self-report measure of executive functions/self-regulation in an everyday environment. It includes 75 items with nine overlapping clinical scales including inhibit, self-monitor, plan/organize, shift, initiate, task monitor, emotional control, working memory, and organization of materials. All items are rated in terms of frequency on a 3-point scale (0 = never, 1 = sometimes, 2 = often). Raw scores for each scale are summed for an overall summary score - the Global Executive Composite (GEC) - and T scores (mean = 50, standard deviation = 10) are determined. Lower scores indicate better executive function. Raw scores are presented here on a scale from 0-150.
Time Frame: Baseline and Week 6
Population: Intent-to-Treat (ITT) Population: all subjects who were randomized and were not an extreme outlier for PERMP-C at Week 6.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 89 | 94
score on a scale | -11.5 (2.19) | -15.6 (2.11)

4. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS)
Description: The HADS consists of 14 items, divided into two 7 item subscales: anxiety (HADS-A) and depression (HADS-D). HADS-A questions reflect a state of generalized anxiety and HADS-D focuses on the concept of anhedonia. Subjects will rate each of the questions on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). Scores will be derived by summing responses for each of the two subscales or for the scale as a whole, and the total score is out of 42, with higher scores indicating higher symptom severity. The HADS-A subscale, scored on a scale from 0-21, will be used in the statistical analysis and presented here.
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 89 | 94
score on a scale | -1.6 (0.38) | -1.9 (0.37)

5. Secondary Outcome: Change From Baseline in Adult ADHD Quality of Life Scale (AAQoL)
Description: The AAQoL is a 29-item self-reported scale evaluating aspects of quality of life in ADHD patients. It consists of a total score of 4 subscales, including life productivity, psychological health, life outlook, and relationship. Items are scored on a 5-point scale ranging from 1 (not at all/never) to 5 (extremely/very often). Raw scores are transformed to a 0 to 100 scale with higher scores indicating a better quality of life.
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 90 | 94
score on a scale | 10.8 (1.53) | 8.4 (1.47)

6. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity (CGI-S)
Description: The CGI-S is a brief assessment tool that measures clinician's impression of illness severity. Evaluation includes information from the subject and may include information from the subject's medical history, physical exam, or other ratings done at screening. CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill). Lower scores indicate less severe symptoms.
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 89 | 95
score on a scale | -0.9 (0.10) | -0.8 (0.10)

7. Secondary Outcome: Responder Rate
Description: Responder rate is defined as the proportion of subjects with ≥ 20-point improvement on PERMP-C or ≥ 2-point improvement on CGI-S from Baseline to Week 6.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 81 | 89
percentage of responders | 64.2 | 60.7

8. Secondary Outcome: Change From Baseline in the ADHD Investigator Symptom Rating Scale - Expanded Version (AISRS-EV)
Description: The expanded version of AISRS includes the 18 items of AISRS plus 13 additional items evaluating executive function deficits and emotional dyscontrol. AISRS-EV items are scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with a total score ranging from 0 to 93. Lower scores indicate less severe symptoms
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NRCT-101SR | Placebo
Number analyzed (Participants) | 89 | 95
score on a scale | -17.1 (1.77) | -15.4 (1.72)

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to approximately Week 7
Description: Safety Population consisted of all participants who received at least 1 dose of study drug. Subjects were analyzed as treated. In the case that a subject was misallocated study drug, they were grouped with active subjects as long as they received any active drug. Data for safety is reported by treatment group (NRCT-101SR and placebo).
Arm/Group | NRCT-101SR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/114
Other Adverse Events (participants affected / at risk) | 42/108 | 36/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NRCT-101SR (N=108) | Placebo (N=114)
Upper respiratory tract infection (Infections and infestations) | 3 | 4
COVID-19 (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 3 | 0
Headache (Nervous system disorders) | 10 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Agitation (Psychiatric disorders) | 3 | 0
Fatigue (General disorders) | 4 | 9
Urinary tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Sedation (Nervous system disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Initial insomnia (Psychiatric disorders) | 1 | 1
Irritability (Psychiatric disorders) | 1 | 1
Anger (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Poor quality sleep (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Terminal insomnia (Psychiatric disorders) | 0 | 1
Pre-existing condition improved (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 2
Dry eye (Eye disorders) | 0 | 1
Weight increased (Investigations) | 1 | 1
Flushing (Vascular disorders) | 1 | 0
Orthostatic hypertension (Vascular disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This agreement establishes that all protocol information, data, and materials related to Neurocentria's study are confidential and Neurocentria's property. Institution retains ownership of subject medical records but must maintain strict confidentiality, sharing information only with necessary parties bound by the same confidentiality terms. Exceptions include publicly available information, third-party disclosures, previously known information, or independently developed information.

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT05683249/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT05683249/SAP_001.pdf